CLINICAL TRIAL: NCT05607225
Title: Deep Learning-based Classification and Prediction of Radiation Dermatitis in Head and Neck
Brief Title: Deep Learning-based Classification and Prediction of Radiation Dermatitis in Head and Neck Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, YE ZHANG, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: JS2022-62
Record Dates: First submitted 2022-10-24; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Radiation Dermatitis; Head and Neck Cancer
MeSH Terms: conditions — Radiodermatitis; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to develop a deep learning-based model to grade the severity of radiation dermatitis (RD) and predict the severity of radiation dermatitis in patients with head and neck cancer undergoing radiotherapy, so as to provide support for doctors' diagnosis and prediction.

DETAILED DESCRIPTION:
1. Image acquisition The images of the neck area were collected from the enrolled patients one week before and every week during radiotherapy. The photographs were taken from three angles (front, left and right oblique) of the neck area.
2. Grading evaluation Each image was individually graded by three experienced radiotherapy experts according to the RD criteria of RTOG
3. Data analysis Construct a dermatitis grading model basing on deep learning. Evaluate the performance of model using accuracy, precision, recall, F1-measure, dice value.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Histologically or cytologically confirmed head and neck carcinoma confirmed by pathology.
* Receive radical radiotherapy including neck area
* Informed consent.

Exclusion Criteria:

* unable to cooperate with image acquisition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with head and neck cancer who will receive radical radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy | July 1, 2022 to June 30, 2025
  Evaluate the rate of deep learning based rating model in accordance with experts' assessment.
Precision | July 1, 2022 to June 30, 2025
  The proportion of positive samples in the positive prediction result
Recall | July 1, 2022 to June 30, 2025
  The proportion of positive samples that were predicted to be positive
F1-measure | July 1, 2022 to June 30, 2025
  The harmonic average of precision and recall
ROC curve | July 1, 2022 to June 30, 2025

SECONDARY OUTCOMES:
dice value | July 1, 2022 to June 30, 2025
  Ratio of overlap and distance between artificial and automatic neck segmentation regions

CONTACTS AND LOCATIONS:
Overall Officials: Ye Zhang, MD, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College; Li Ma, MD, Principal Investigator — Shenzhen Cancer Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Shenzhen Cancer Hospital, Chinese Academy of Medical Sciences, Shenzhen, Guangdong
  - Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College, Beijing

IPD SHARING:
Plan to Share IPD: No